CLINICAL TRIAL: NCT00006245
Title: Phase II Trial of Flavopiridol and Paclitaxel in Patients With Paclitaxel-Refractory Esophageal Cancer
Brief Title: Flavopiridol and Paclitaxel in Treating Patients With Locally Advanced or Metastatic Esophageal Cancer That Has Not Responded to Previous Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068176; MSKCC-00060; NCI-1672
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Esophageal Cancer
Keywords: stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — alvocidib; Paclitaxel

INTERVENTIONS:
Drug: alvocidib
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining flavopiridol and paclitaxel in treating patients who have locally advanced or metastatic esophageal cancer that has not responded to previous paclitaxel therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with paclitaxel-refractory locally advanced or metastatic esophageal cancer treated with sequential paclitaxel and flavopiridol.
* Determine the toxicity of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.
* Obtain pharmacokinetic information about this regimen.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours on day 1 and flavopiridol IV continuously over 24 hours on day 2 weekly for 3 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, after courses 1 and 2, and then every 2 courses thereafter.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 6-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or carcinoma of the gastroesophageal (GE) junction

  * If tumor extends below the GE junction into the proximal stomach, 50% of the tumor must involve the esophagus or GE junction
  * No gastric cancers with only a minor involvement of the GE junction or distal esophagus
* Metastatic or locally advanced disease that is considered surgically unresectable
* Must have failed a prior chemotherapy regimen that included paclitaxel for metastatic disease OR
* Failed prior combination taxane-based chemotherapy and radiotherapy for locally advanced disease

  * Must have documented evidence of the following:

    * Disease progression while on taxane-based neoadjuvant or adjuvant therapy OR
    * Recurrent disease within 6 months of therapy
* Measurable disease

  * Accurately measured in at least 1 dimension

    * At least 20 mm by conventional techniques OR
    * At least 10 mm by spiral CT scan
  * The following are considered nonmeasurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusions
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No active angina or myocardial infarction within the past 6 months
* No significant ventricular arrhythmia requiring antiarrhythmic medication
* Atrial fibrillation that is well controlled on standard management allowed

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study
* No preexisting peripheral neuropathy of grade 2 or greater
* No serious concurrent infection
* No uncontrolled, nonmalignant medical illness that would preclude study
* HIV negative
* No other active malignancy within the past 5 years except:
* Nonmelanoma skin cancer or
* Carcinoma in situ of the cervix
* History of T1a or T1b prostate cancer (detected incidentally during transurethral resection of the prostate and comprising less than 5% of resected tissue) allowed if PSA normal since surgery
* No medical or psychiatric condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* No more than 6 months since prior paclitaxel
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed (indicator lesion must be outside of prior radiation port unless recent evidence of disease progression at that site)
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No prior cyclin-dependent kinase or protein kinase C inhibitors for esophageal cancer
* Recovered from toxic effects of any prior therapy
* No concurrent vitamins, antioxidants or herbal preparations or supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Rathkopf DE, Ilson DH, Yi S, et al.: A phase II trial of sequential paclitaxel and flavopiridol in patients with metastatic paclitaxel-refractory esophageal cancer. [Abstract] American Society of Clinical Oncology 2004 Gastrointestinal Cancers Symposium, 22-24 January 2004, San Francisco, CA. A-67, 2004.